CLINICAL TRIAL: NCT03516929
Title: Non-selective Assessment of Carotid Artery Stenosis and Lower Limb Peripheral Ischemia Prior to Coronary Artery Bypass Surgery
Brief Title: Assessment of Carotid Artery Stenosis and Lower Limb Peripheral Ischemia Prior to CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mr Ihab Ali (Other)
Responsible Party: Sponsor-Investigator, Mr Ihab Ali, Assistant Professor of Cardio-thoracic Surgery at Ain-Shams University, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 25/2018
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Carotid Artery Diseases; Peripheral Artery Disease
Keywords: carotid; peripheral arterial disease; endarterectomy
MeSH Terms: conditions — Carotid Artery Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high risk group (Active Comparator): history of stroke or TIA, carotid bruit, left main stem disease, other peripheral vascular disease
  Interventions: Diagnostic Test: carotid duplex, both LL arterial duplex
- low risk group (Sham Comparator): No history or stroke,TIA. NO left main stem disease
  Interventions: Diagnostic Test: carotid duplex, both LL arterial duplex

INTERVENTIONS:
Diagnostic Test: carotid duplex, both LL arterial duplex — assessment of carotid stenosis and lower limb peripheral ischemia.

SUMMARY:
From our experience among Egyptian population in our institution, there is an increased prevalence of hidden subclinical peripheral artery disease along with carotid artery affection. Thus, increasing the risk of post-operative morbid complications.We aim to evaluate routine/ non-selective carotid and peripheral arterial screening in asymptomatic patients undergoing coronary artery bypass grafting in the Egyptian populationIt is a prospective, non-randomized, comparative study including two groups of patients. The study will start from the day of approval of the ethical committee. It will include 260 patients, on basis of "all new comers". Patients will be examined and classified as "high-risk" group (ɳ = 130) or "low-risk" group (ɳ=130).

All patients will have the "routine" preoperative investigations along with evaluation of extracranial carotid system by non-invasive carotid duplex and lower limb arterial system by non-invasive bilateral lower limb arterial duplex.

ELIGIBILITY:
Inclusion Criteria:

1. The acceptance of the patients to participate in the study in the form of a written consent.
2. Patients of both sexes.
3. Three vessels disease for CABG.
4. Patients' age: from 35 to 75 years old.
5. Elective, isolated, primary cases of CABG.
6. Patients with ejection fraction above 40%.
7. Inclusion criteria for the high-risk group will include:

   1. Patients with preoperative history of cerebrovascular events or symptoms suggestive of CVS eg.TIA, transient blindness in one eye, Dizziness, Confusion, Drowsiness, Headache, Temporary inability to speak or move.
   2. Carotid bruit
   3. Left main stem coronary artery disease
   4. Presence of other peripheral vascular disease

Exclusion Criteria:

1. Patients refusing to participate in the study.
2. Age 76 years or above
3. Morbid obese patients (body mass index more than 35).
4. Patients who underwent coronary stenting before.
5. Patients who underwent previous cardiac operation before.
6. Patients with impaired renal functions (serum creatinine > 1.5 mg/dl, blood urea > 100 mg/dl and K+ > 5 meq/L).
7. Patients with preoperative hemoglobin < 9 gm/dl, white blood cells > 15,000 cells/mcl,platelets count < 140,000 per microliter.
8. Patients with rhythm defects by electrocardiography (ECG).
9. Patients with preoperative O2 saturation < 90 % by pulse oximetry.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
culprit pathology in carotid and / or lower limb duplex | 6 months

SECONDARY OUTCOMES:
new cerebrovascular event or lower limb ischemia in the post operative period | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio-thoracic Academy -Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali I, Shokri H, Abd Al Jawad M. Assessment of carotid artery stenosis and lower limb peripheral ischemia before coronary artery bypass grafting operations: a non-randomized clinical trial. J Cardiothorac Surg. 2020 Sep 29;15(1):283. doi: 10.1186/s13019-020-01340-7. PMID 32993716